CLINICAL TRIAL: NCT06867497
Title: A Multi-center, Open-label, Randomized, Two-stage, Two-way Crossover Bioequivalence Study to Compare and Evaluate the Pharmacokinetic Characteristics and the Safety Between Administration of BR2021 and BR2021-1 in Patients With Metastatic Adenocarcinoma of the Pancreas
Brief Title: A Study to Compare and Evaluate the Pharmacokinetic Characteristics and the Safety Between Administration of BR2021 and BR2021-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-ABX-CT-101
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Adenocarcinoma of the Pancreas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test drug (Experimental)
  Interventions: Drug: BR2021
- Reference drug (Active Comparator)
  Interventions: Drug: BR2021-1

INTERVENTIONS:
Drug: BR2021 — intravenous administration for 30 minutes
  Arms: Test drug
Drug: BR2021-1 — intravenous administration for 30 minutes
  Arms: Reference drug

SUMMARY:
The purpose of this clinical study is to compare and evaluate the pharmacokinetic characteristics and the safety between administration of BR2021 and BR2021-1 in patients with metastatic adenocarcinoma of the pancreas

ELIGIBILITY:
Inclusion Criteria:

* Those with histologically or cytologically proven metastatic adenocarcinoma of the pancreas
* Those who agree to rule out the possibility of their and their spouses' or sexual partners' pregnancy by using medically recognized methods of contraception (contraceptives administration & transplantation or intrauterine device(IUD), sterilization(vasectomy, tubal ligation, etc.), barrier methods (spermicide & male condom, combined use of contraceptive diaphragm, sponge or cervical cap)) from the date of the first administration of the investigational products to at least 6 months after the last administration date and disagree to provide their sperm or ovum.
* Those who spontaneously decide to participate and sign written consent to comply with the subject's precautions after listening to and fully understanding detailed explanation of this clinical trial

Exclusion Criteria:

* In the case of a female subject, pregnant woman or those suspected pregnancy or lactating woman.
* Those who have to administer this study's contraindicated drugs with the investigational product from 2 weeks before the participation until end of this study
* Those who can't discontinue a diet (ex. raw grapefruit, grapefruit juice or food containing grapefruit, etc.) that may affect the absorption, distribution, metabolism, and excretion of the drug from 48 hours before the first administration date to post study visit(PSV)
* Those who can't discontinue other drugs except the investigational product of this study that may affect the metabolism and excretion of the drug for the entire study period (However, if necessary, such as treatment of adverse event, it can be administrated according to investigator's judgment)
* Those who have participated in other clinical trials(including bioequivalence tests) and administered their investigational products within 4 weeks before the first administration date (However, the termination for participation in other clinical trials are based on the last administration date of their investigational products) or those whose last administration date of their investigational products of other clinical trials doesn't elapse five times the half-life of their investigational products based on the first administration date of investigational product of this study

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-10-28 (Estimated); Study Completion 2025-10-28 (Estimated)

PRIMARY OUTCOMES:
AUCt | 0~72 hours after administration
  Area under the Plasma Concentration-Time Curve from 0 to time t
Cmax | 0~72 hours after administration
  Maximum Concentration of Drug in Plasma

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No